CLINICAL TRIAL: NCT07107074
Title: A Phase 2b, Multicenter, Randomized, Placebocontrolled, Double-blind Study to Assess the Safety and Efficacy of AD04 in Patients With Early Alzheimer's Disease - ADVANCE
Brief Title: Effects of a Widely Used Vaccine Adjuvant in Subjects With Early Alzheimer's Disease Double-blind Study to Assess the Safety and Efficacy of AD04 in Patients With Early Alzheimer's Disease - ADVANCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ADvantage Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADVANCE-AD04-001
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1ml AD04 (Experimental): Each patient will receive 6 single s.c. injections of IMP at monthly intervals over a 5-month treatment period.
  Interventions: Drug: AD04
- 1ml PBS (Placebo Comparator): Each patient will receive 6 single s.c. injections of placebo at monthly intervals over a 5-month treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD04 — Each patient will receive 6 single s.c. injections of IMP at monthly intervals over a 5-month treatment period.
  Arms: 1ml AD04
Drug: Placebo — Each patient will receive 6 single s.c. injections of Placebo at monthly intervals over a 5-month treatment period.
  Arms: 1ml PBS

SUMMARY:
The purpose of this randomized, placebo-controlled phase 2b study is to prospectively evaluate AD04's potential as a disease-modifying drug in AD. By evaluating the safety, pharmacodynamics, and efficacy of AD04 in early AD patients, we aim to deliver a comprehensive and robust data set that furthers our understanding of the effects of AD04 in AD pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-85 years old
2. Has a diagnosis of probable AD based on the National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, integrating both clinical and neuropathological criteria
3. Has a Mini-Mental State Examination (MMSE) score between 22 and 30. Note: Regarding inclusion criterion #2, it is obvious that patients with an MMSE score ≥27 may not fulfill all NINCDS/ADRDA criteria, especially those referring to or requiring a state of dementia. In such cases, inclusion criteria #4 and #5 ensure the specificity of the diagnosis (prodromal stage of AD/AD-type mild cognitive impairment [MCI]).
4. Has brain MRI showing medial temporal lobe atrophy as assessed by the Scheltens' scale (score ≥2, at least at one site) or has AD-type CSF signature at a 7:3 ratio of Scheltens to CSF signature. This criterion was chosen with the goal of having a patient cohort which reflects as closely as possible that of the AFF006 study; specific cut-offs for CSF AD biomarkers will be defined based on the methodology of the selected central laboratory.
5. Has a Free and Cued Selective Reminding Test (FCSRT) total recall ≤40 or free recall ≤17, indicating hippocampal damage, episodic memory impairment, and amnestic syndrome
6. Must have results of a physical examination, including visual and auditory acuity within the acceptable range for the age group to allow neuropsychological testing
7. Has Hachinski Ischemia Scale score ≤4 to distinguish AD from vascular dementia
8. Written informed consent of study-related procedures and of genetic investigations signed and dated by the patient and the caregiver
9. Availability of a partner/caregiver knowing the patient and being able to accompany the patient at the visits. He/ she will be in frequent contact with the participant (defined as at least 10 hours per week), will accompany the participant to the planned study visits and/or be available by telephone at designated times
10. Women of childbearing potential and men with female partners of childbearing potential must use 2 effective methods of birth control during the course of the trial and for at least 90 days after the last dose in a manner such that risk of failure is minimized. Male participants should refrain from donating sperm during the intervention period and for at least 90 days after the last dose of study intervention

    Exclusion Criteria:
    * Known or suspected allergy, or history of anaphylaxis, to vaccines or their excipients, if considered relevant by the Investigator
    * Any medical or neurological condition (other than AD) that might cause the participant's cognitive impairment, including:
    * History or evidence of cerebrovascular disease (stroke, transient ischemic attack, intracerebral hemorrhage), or diagnosis of possible, probable or definite vascular dementia in accordance with National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN) criteria
    * A significant number of >4 microhemorrhages, a single prior hemorrhage > 1 cm3, >2 lacunar infarcts, a single prior infarct > 1 cm3, radiological finding supporting the NINDS-AIREN criteria as operationalized in Stroke. 2003 Aug;34(8):1907-12, meningioma with a perpendicular diameter of >1cm or significant mass effect on the brain parenchyma, evidence of a cerebral contusion, encephalomalacia, aneurysms, brain neoplasms such as gliomas or subdural hematoma/effusion with a diameter of >1cm, diffuse white matter disease (Fazekas score - deep white matter score >3) or significant mass effect on the brain parenchyma assessed by MRI at screening
    * Evidence of a clinically relevant Parkinson's disease, dementia with Lewy bodies, frontotemporal dementia, progressive supranuclear palsy, corticobasal degeneration, amyotrophic lateral sclerosis, Huntington's disease, multiple sclerosis, mental retardation, hypoxic cerebral damage, or head trauma with loss of consciousness that led to persistent cognitive deficits
    * Refractory epilepsy (has had seizures within the past 2 years)
    * Has had a history within the last 5 years of a serious infectious disease affecting the brain
    * Clinically significant unstable psychiatric illness in the past 6 months
    * Has a Geriatric Depression Scale score > 6 (on the staffadministered short form)
    * Hypothyroidism or vitamin B12 deficiency (patients with corrected hypothyroidism or vitamin B12 deficiency are eligible for the study provided that treatment has been stable for 3 months before study entry)
    * Patients with long covid-19 showing long-term neurological sequelae within the past 12 months at the time of screening
    * History of chronic alcohol or drug abuse/ dependence within the past 5 years
    * Patient with past or present suicidal ideation and intent as assessed by the Columbia Suicidality Severity Rating Scale (CSSRS), or who, in the clinical judgment of the investigator, presents a serious risk of suicide
    * Presence of autoimmune disease, autoinflammatory syndrome, or immunological deficiency syndrome (including human immunodeficiency virus (HIV) infection)
    * Relevant cardiovascular, hepatic, gastroenterological, respiratory, endocrinological, hematologic disease, or any other condition that, in the Investigator's opinion, could interfere with the analyses of safety and efficacy in this study, unless patient has been on stable doses of medication for any of these concurrent illnesses for at least 3 months prior to study entry
    * History within the last 2 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen posttreatment; or has a life expectancy of <2 years.
    * Presence of end stage kidney failure (on dialysis) (which may affect renal clearance of aluminium)
    * Patient has hemochromatosis
    * If on conventional AD therapies such as donepezil or memantine, anticholinergics in general (including neuroleptics with anticholinergic properties, certain bladder relaxants, anticholinergic drugs for use in lung diseases), or lipid-modifying therapies, doses must be stable for at least 3 months prior to the screening visit and during the entire trial period
    * Current or anticipated use of immunosuppressive drugs such as, but not limited to, azathioprine, cyclosporine, methotrexate, tacrolimus, or mycophenylate within 2 months or any myelosuppressive or cytotoxic chemotherapies within the 12 months prior to the screening visit. Use of systemic corticosteroids equivalent to ≥20mg/week prednisone within the past 4 weeks before screening and during the course of the study (intranasal or inhaled steroids for allergies/asthma is allowed)
    * Current or anticipated use of allergy immunotherapies
    * Patient has received or plans to receive any aluminium-adjuvanted vaccines within 14 days prior to any dose of study drug
    * Pregnancy
    * Contraindication for MRI imaging, including but not limited to pacemakers; cochlear implants, cerebral aneurysm clips; implanted infusion pumps; implanted nerve stimulators; metallic splinters in the eye; other magnetic, electronic, or mechanical implants; claustrophobia; inability to lie motionless for 30 minutes; or any other clinical history or examination finding that, in the judgement of the Investigator, would pose a potential hazard in combination with MRI
    * Contraindication for CSF collection, including certain conditions and / or medications such as high doses of blood thinning agents
    * Patient has received any vaccine targeting Aβ or tau for the treatment of AD. For all other experimental AD drugs, including passive immunotherapies, participation in the active treatment phase of any AD clinical trial within 3 months (or 5 half-lives, whichever is longer), prior to Visit 1
    * Participation in the active treatment phase of any non-AD clinical trial within 30 days prior to Visit 1
    * Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the Sponsor

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Composite score assessing cognition (aADAS-cog), daily function Activities of Daily Living (aADCS-ADL) and a global dementia severity score (CDR-sb) over 6 months measured in overall time saved with treatment | 6 months
  Based on the evaluation of the time savings in cognitive, functional and global domains.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 12 months
Change from baseline in Clinical Dementia Rating - sum of boxes (CDRsb) | 12 months
Change from baseline in hippocampal volume (total, right, and left), measured by volumetric Magnetic Resonance Imaging (MRI) | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Achim Schneeberger, MD, Study Director — ADvantage Therapeutics
Locations (3):
- Institute Neuromed, Korneuburg, Lower Austria, Austria
- Poland (2):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Promente-Centrum Neurologii i Psychogeriatrii, Bydgoszcz

IPD SHARING:
Plan to Share IPD: No